CLINICAL TRIAL: NCT05694182
Title: The Safety and Efficacy of an Oral Superfruits Supplement for Skin Brightening and Wrinkle Reduction
Brief Title: The Safety and Efficacy of an Oral Superfruits Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMRAMREC003-22
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral superfruits supplement (Experimental): Participants will consume oral superfruits supplement once daily for 6 weeks.
  Interventions: Other: Other: Oral superfruits supplement

INTERVENTIONS:
Other: Other: Oral superfruits supplement — The supplement contain superfruits that are beneficial for human health

SUMMARY:
This study is conducted to evaluate the safety and effectiveness of an oral superfruits supplement for skin brightening and wrinkle reduction. Superfruits are reported to have high bioactive compounds with beneficial effects on human health. The study duration is 12 weeks and the skin assessment will be carried out at baseline, week 2, week 6 and week 12. The participants will consume the supplement for 6 weeks and at week 12, final skin assessment will be conducted. The main questions this study aims to answer are:

1. The skin brightening effect of the oral superfruits supplement.
2. The effect of the oral superfruits supplement on wrinkle reduction.
3. To observe any adverse effect occurrence with the consumption of the oral superfruits supplement.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian citizen
* Male and female (age 20-60 years old)

Exclusion Criteria:

* Participant who taking any dietary supplements for the past 4 weeks which can affect the study results
* Participant who are on contraceptive pills for the past 3 months
* Participant who undergo cosmetics treatments such as botox, filler and laser and light treatment within the last 3 months
* Pregnant or plans to get pregnant and breastfeeding women

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in skin tone from baseline and at week 2, week 6 and week 12 after consumption of the superfruits supplement | Baseline, week 2, week 6 and week 12
  Skin tone will be assessed using JANUS III skin analyzer
Changes in skin wrinkles from baseline and at week 2, week 6 and week 12 after consumption of the superfruits supplement | Baseline, week 2, week 6 and week 12
  Skin wrinkles will be assessed using JANUS III skin analyzer and Wrinkle Severity Rating Scale (WSRS). For WSRS, dermatologists will evaluate participants' wrinkles based on 5-point photonumeric rating scale that will objectively evaluate the severity of crow's feet at rest (static) and with a smiling expression (dynamic). The scale scores are 0 for no wrinkles, 1 for very fine wrinkles, 2 for fine wrinkles, 3 for moderate wrinkles, and 4 for severe wrinkles.
Adverse effect after consumption of the superfruits supplement | Week 12
  Based on adverse effect occurrence on participants that occur during study period (12 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No